CLINICAL TRIAL: NCT07116018
Title: Feasibility Testing of an Adapted Psychoeducational Intervention for Caregivers of Patients Undergoing Allogeneic Stem Cell Transplant for Hematological Malignancy
Brief Title: Psychoeducation for AlloHCT Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Samantha Mayo, Clinician Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-5539
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Caregivers; Stem Cell Transplant; Psychoeduction; Coping
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychoeducational intervention (Experimental): The intervention will be psychoeducational program, comprising a series of 8 individual sessions over a 12 week period. The intervention is a manualized, adapted version of the Psychoeducation, Paced Respiration, and Relaxation (PEPRR) intervention (Laudenslager et al. 2015).
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — The intervention comprises 8 individual psychoeducational sessions over 12 weeks, as an adaptation of the Psychoeducation, Paced Respiration, and Relaxation (PEPRR) (Laudenslager et al., 2015). The adaptation in the current study involves delivery by a trained nurse and omission of the biofeedback component.

SUMMARY:
Background: Caregivers of patients undergoing allogeneic hematopoietic cell transplantation (alloHCT) for hematological malignancies face significant challenges that can impact their well-being. This study aims to evaluate the feasibility and acceptability of an adapted psychoeducational intervention(PEI) designed to support these caregivers.

Methods: This study will recruit caregivers of alloHCT patients. Participants will be enrolled during pre-transplant clinic visits, typically 2-4 weeks before the scheduled transplant. The intervention consists of eight sessions over 12 weeks, delivered via Microsoft Teams by a nurse facilitator. In the adapted PEI, participants will learn stress management, coping strategies, energy management, goal-setting, communication skills, and support resource access through interactive exercises. Data Collection: Participants will complete questionnaires at three time points: pre-intervention, one month post-transplant, and three months post-transplant. The final assessment will include additional questions about feasibility, acceptability and the initial efficacy of the adapted PEI.

Outcomes: The primary outcomes will be the feasibility and acceptability of the adapted psychoeducational intervention (PEI). Secondary outcomes will include initial efficacy of the adapted PEI on caregiver outcomes such as depression, anxiety, satisfaction with caregiving and quality of life.

Significance: This research aims to assess the feasibility, acceptability and initial efficacy of implementing the adapted PEI for alloHCT caregivers. If found feasible and acceptable, this intervention could potentially improve caregivers' ability to manage caregiving stressors and pave the way for larger-scale randomized studies and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Must be caregiver for an adult patient diagnosed with hematological malignancy who is scheduled to receive allogeneic stem cell transplant.
* Are recruited and consented to participate in the caregiver study during the patient's pre-transplant screening phase for allogeneic stem cell transplant.
* Will provide care for the patient from the day of allogeneic stem cell transplant up to 100 days post- transplant.
* Are willing to begin the study intervention no earlier than 0-day post-transplant and not later than 2-weeks post-transplant.

Exclusion Criteria:

* Less than 18 years of age
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | 3 months
  The Feasibility of Intervention Measure (FIM) revised to evaluated the psychoeducation program comprises 4-items regarding the respondent's perceptions of the feasibility of the intervention. Responses range from 1 (completely disagree) to 5 (completely agree). Scale value is computed by averaging responses and ranges from 1-5. Higher values indicate greater feasibility of the intervention.
Acceptability of Intervention Measure (AIM) | 3 months
  The Acceptability of Intervention Measure (AIM) revised to evaluated the psychoeducation program comprises 4-items regarding the respondent's perceptions of the acceptability of the intervention. Responses range from 1 (completely disagree) to 5 (completely agree). Scale value is computed by averaging responses and ranges from 1-5. Higher values indicate greater acceptability of the intervention.
Intervention Appropriateness Measure (IAM) | 3 months
  The Intervention Appropriate Measure (IAM) revised to evaluated the psychoeducation program comprises 4-items regarding the respondent's perceptions of the appropriateness of the intervention. Responses range from 1 (completely disagree) to 5 (completely agree). Scale value is computed by averaging responses and ranges from 1-5. Higher values indicate greater appropriateness of the intervention.

SECONDARY OUTCOMES:
Perceived Stress | Baseline, 1 month, 3 months
  Perceived Stress Scale (PSS)
Depression | Baseline, 1 month, 3 months
  Centre for Epidemiological Studies- Depression (CES-D) scale
Caregiver Quality of Life | Baseline, 1 month, 3 months
  Caregiver Quality of Life Index- Cancer Scale
Satisfaction with Life | Baseline, 1 month, 3 months
  Satisfaction with Life Scale
Anxiety | Baseline, 1 month, 3 months
  State-Trait Anxiety Inventory (STAI)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Mayo, RN, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laudenslager ML, Simoneau TL, Kilbourn K, Natvig C, Philips S, Spradley J, Benitez P, McSweeney P, Mikulich-Gilbertson SK. A randomized control trial of a psychosocial intervention for caregivers of allogeneic hematopoietic stem cell transplant patients: effects on distress. Bone Marrow Transplant. 2015 Aug;50(8):1110-8. doi: 10.1038/bmt.2015.104. Epub 2015 May 11. PMID 25961767